CLINICAL TRIAL: NCT02689297
Title: Three Different Oral Hygiene Regimes on Three Volatile Sulfur Compounds
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tokyo Medical and Dental University (Other)
Responsible Party: Principal Investigator, Ei Ei Aung, Graduate student, Department of Oral Health Promotion, Tokyo Medical and Dental University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OHP-018-EI-2
Record Dates: First submitted 2016-02-08; First posted 2016-02-23 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Halitosis
MeSH Terms: conditions — Halitosis | interventions — chlorine dioxide

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- group A (Other): Mouthwash (chlorine dioxide 12ml two times per day, for three weeks)
  Interventions: Other: chlorine dioxide
- group B (Other): Small toothbrush for tongue cleaning two times per day for three weeks
  Interventions: Other: small toothbrush for tongue cleaning

INTERVENTIONS:
Other: chlorine dioxide — First week, subjects were instructed to do regular tooth brushing. After that group A was requested to use chlorine dioxide mouthwash two time per days for three weeks in addition to tooth brushing and then, one week for combination of tooth brushing, tongue cleaning and mouth washing.
  Arms: group A
Other: small toothbrush for tongue cleaning — First week, subjects were instructed to do regular tooth brushing. After that group B was requested to brush their tongue with small toothbrush two time per days for three weeks in addition to tooth brushing and then, one week for combination of tooth brushing, tongue cleaning and mouth washing.
  Arms: group B

SUMMARY:
The purpose of the study is to evaluate the effect of various oral hygiene regimes on three volatile sulfur compounds.

DETAILED DESCRIPTION:
Thirty male monk volunteers who matched with the including criteria were divided randomly into two groups. Both groups were practiced to brush their teeth with scrubbing method for one week. Then, each group were instructed to do different additional protocol regimen- group A have to do mouth washing and tooth brushing and group B have to practice tongue cleaning addition to tooth brushing for three weeks. At the fifth week, both groups were instructed to practice tooth brushing, mouth washing and tongue cleaning. Three different volatile sulfur compounds were measured by oral chroma. Tongue characteristics, oral examination were checked as the outcomes of this study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of oral malodor
* No systemic diseases and no severe dental diseases
* At least 20 functional teeth

Exclusion Criteria:

* Risky oral habit (smoking and betel quid chewing)
* Current use of antibiotics or any drugs
* Current use of any kind of mouthwash

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Three different volatile sulfur compounds | up to 5weeks
  Investigator measured three different volatile sulfur compounds: hydrogen sulfide, methyl mercaptan, dimethyl sulfide concentrations (ng/10ml) by using Oral chroma.

SECONDARY OUTCOMES:
Oral Health examination | up to 5weeks
  As oral examination, investigator examined present teeth, DMF-T (decayed, missing and filled teeth)
Tongue coating characteristics | up to 5weeks
  As tongue coating characteristics, investigator examined tongue coating score (by using winkle tongue coating index) at the baseline, one week later, four weeks later and five weeks later.
Number of teeth with bleeding on probing | up to 5weeks
Plaque index score | up to 5weeks